CLINICAL TRIAL: NCT05211843
Title: Saliva Insulin as Biomarker of Risk Factors for Metabolic Dysregulation and Caries Which Can be Limited by Drinking Water Intervention in Elementary School Age Children
Brief Title: Saliva Insulin as Biomarker of Risk Factors for Metabolic Dysregulation and Caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jodi Stookey (Other Government)
Responsible Party: Sponsor-Investigator, Jodi Stookey, MCAH Senior Epidemiologist, San Francisco Department of Public Health
Organization: San Francisco Department of Public Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Saliva insulin biomarker
Record Dates: First submitted 2021-12-17; First posted 2022-01-27 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Caries; Metabolomic Profile
MeSH Terms: interventions — Drinking Water

STUDY DESIGN:
Intervention Model Description: Three randomly assigned groups, with randomization stratified by weight status, with measurements at baseline and post-intervention
Who Masked: Outcomes Assessor
Masking Description: The participant will know what group they are assigned to as they will see and taste the assigned beverage. The investigator who assigns participants to a treatment group will not administer the beverage or collect data. The investigator who administers the beverage will know the group assignment. The laboratory staff who assess the outcomes will not know the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No drink (No Intervention): Control; Participants will receive no drink
- Drinking water (Experimental): Intervention drink; Participants will receive 500 ml drinking water from the San Francisco tap (i.e. fluoridated tap water). 500 ml is the standard bottle size.
  Interventions: Other: Drinking water
- Apple juice (Active Comparator): Intervention drink; Participants will receive 200 ml box of apple juice. 200 ml is the standard serving usually available to this study population in the school setting
  Interventions: Other: Apple juice

INTERVENTIONS:
Other: Drinking water — The intervention will compare the effects of a usual serving of drinking water with the effects of a usual serving of apple juice. Both beverages will also be assessed relative to the effects of not drinking anything at all.
  Arms: Drinking water
Other: Apple juice — apple juice
  Arms: Apple juice

SUMMARY:
Saliva insulin shows promise as a non-invasive biomarker of high carbohydrate intake and/or insulin resistance, key risk factors for metabolic dysregulation and caries.

Saliva insulin monitoring could potentially inform the planning and evaluation of interventions to prevent child obesity, diabetes and caries, without relying on self-reported measures from children, parents, child care providers or teachers.

School-based public health screening programs, which have staff and data collection infrastructure in place to regularly and systematically collect saliva during oral health screening, have opportunity to monitor saliva insulin.

This randomized controlled trial explores if saliva insulin is responsive to the kinds of obesity and caries intervention currently in progress in schools, namely drinking water intervention. Public health programs may justify adding saliva collection to protocol already in place if saliva insulin data are found to be actionable, i.e. sensitive to risk and intervention.

DETAILED DESCRIPTION:
This randomized controlled trial explores if saliva insulin is responsive to the kinds of obesity and caries intervention currently in progress in schools, namely drinking water intervention.

The specific aims of this randomized controlled trial are to:

Determine if the standard serving (500 ml) of drinking water normalizes saliva insulin to a greater extent, within 60 min, than no beverage or a standard serving (200 ml) apple juice in elementary school age children.

Determine if, in line with lower saliva insulin, 500 ml drinking water significantly alters macronutrient metabolism, within 60 min, relative to no beverage or 200 ml apple juice.

Determine if 500 ml drinking water reduces caries risk factors, improves saliva osmolality, pH, buffering capacity and immune response to a greater extent, within 60 min, than no beverage or 200 ml apple juice.

ELIGIBILITY:
Inclusion Criteria:

UCSF Pediatric Dental Clinic patients New patient exam or recall exams Caregiver and child speak English, Spanish or Chinese Ages 5-10 years San Francisco residents Non-acutely ill (healthy enough to attend school, no fever and no systemic conditions)

Exclusion Criteria:

Child and caregiver do not speak English, Spanish or Chinese Not a San Francisco resident Under age 5 years Over age 10 years Child unwilling to accept randomized drink assignment Child unable or unwilling to drink water or apple juice Child unable or unwilling to give saliva Child is presenting to the dental clinic for an operative procedure Acute illness, fever, infection or condition that would prevent the child from attending school No remaining space in study group (weight-specific recruitment is complete).

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Lower saliva insulin after drinking water compared to juice; compared to no drink | 1 hour
  Lower mean saliva insulin; Greater relative odds of saliva insulin below 5mU/I

SECONDARY OUTCOMES:
Different untargeted metabolomic profile after drinking water compared to juice; and after drinking water compared to no drink | 1 hour
  The metabolomic profile will be measured by Untargeted Profiling of Primary Metabolism by mass spectrometry at the University of California Davis West Coast Metabolomics Center. Metabolomic data analyses will be done on data normalized by creatinine, log transformed, and mean centered using metaboanalyst software. The metabolomic profiles will be evaluated using Orthogonal Partial Least Squares Discriminant Analysis 2-D score plots and Principal Components Analysis score plots. Both types of analyses are required because each has limitations. This study hypothesizes that in both types of analysis, the 95% confidence ellipse for the saliva metabolomic profile after drinking water does not overlap the 95% confidence ellipse for the metabolomic profile after apple juice; nor does it overlap the 95% confidence ellipse after no drink.
Higher saliva pH (potential of hydrogen) after drinking water than after apple juice or no drink | 1 hour
  Mean change in saliva pH from baseline to 1 hour after drinking water is significantly more positive than the mean change in saliva pH after apple juice (anticipating a decrease in saliva pH following the apple juice drink)
Higher saliva buffering capacity after drinking water than after apple juice or no drink | 1 hour
  Greater relative odds of not having 'low' saliva buffering capacity after drinking water compared to apple juice, with 'low' as defined by the CRT buffer capacity test (Ivoclar, Vivadent, Schaan, Liechtenstein); similarly greater odds of not having 'low' buffering capacity after drinking water vs no drink; Greater odds of an improvement in buffering capacity classification (change from baseline to 1 hour after drink treatment) after drinking water compared to apple juice or no drink
Significantly higher saliva secretory immunoglobin a (IgA) after drinking water than after apple juice or no drink | 1 hour
  Mean change in saliva IgA concentration from baseline to 1 hour after drinking water

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Stookey, PhD, Principal Investigator — San Francisco Department of Public Health; Thomas Tanbonliong, DDS, Principal Investigator — University of California, San Francisco; Mimansa Cholera, DDS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Pediatric Dentistry, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No